CLINICAL TRIAL: NCT00063024
Title: Behavioral Strategies to Prevent Osteoporosis in Girls
Brief Title: Program to Prevent Osteoporosis in Girls
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01HD037743 (NIH)
Record Dates: First submitted 2003-06-19; First posted 2003-06-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Osteoporosis
Keywords: Bone health; Weight-bearing physical activity; Calcium
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Behavioral: Increased calcium intake
Behavioral: Weight-bearing physical activity

SUMMARY:
Osteoporosis is a condition defined by decreased bone mass. Osteoporosis generally affects older women and can lead to bone fractures. One way to prevent osteoporosis is to build strong, healthy bones during childhood. This study will evaluate a program designed to improve girls' bones. The program encourages eating foods rich in calcium and participating in physical activity.

DETAILED DESCRIPTION:
Osteoporosis affects more than 25 million people in the United States. The majority of bone fractures in older women are related to osteoporosis. Calcium intake and physical activity are two modifiable behaviors associated with peak bone mass. Interventions targeting these behaviors among youth have tremendous public health potential for preventing osteoporosis. This study will assess the feasibility and effectiveness of a 2-year behavioral program designed to increase calcium intake and physical activity among girls ages 9 to 11.

Thirty Girl Scout troops will be recruited for the study. Girls will be randomized either to the eating and exercise behavior change program or to a control group. Program components focus on behavioral skills development, goal setting, and self-monitoring for dietary calcium intake and physical activity. The program also works to increase social support from peers and parents. The program will take place during 10 weeks of both the 5th and 6th grade years. The program also includes supporting programs during winter and summer breaks. Outcome assessments will be conducted at baseline, and at 6, 12, and 24 months. Primary outcomes will include dietary calcium intake, physical activity, and bone mineral density.

ELIGIBILITY:
Inclusion Criteria

* Member of a Girl Scout troop with at least eight 5th grade girls
* Member of the Greater Minneapolis or St. Croix Valley Girl Scout organization
* Only troops with unanimous parental consent will be included in the trial

Ages: 9 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 322
Dates: Start 1999-06; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Simone A. French, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Division of Epidemiology, School of Public Health, University of Minnesota, Minneapolis, Minnesota, United States